CLINICAL TRIAL: NCT04711525
Title: Interactive Malaysian Childhood Healthy Lifestyle Program (i-MaCHeL) Intervention for Preschool's Child-parent Dyads to Prevent Childhood Obesity: A Cluster-randomized Controlled Trial
Brief Title: i-MaCHeL Study is a Two-group, Cluster-RCT, Involves 460 Preschool's Child-parent Dyads, to Prevent Childhood Obesity
Acronym: i-MaCHeL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sultan Zainal Abidin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UniSZA/UHREC/2020/184
Record Dates: First submitted 2021-01-02; First posted 2021-01-15 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Childhood Obesity Prevention
Keywords: Obesity; Preschool children; Web based program; Body Mass Index; Dietary intake; Physical activity; Health related quality of life; Self efficacy; Role modeling; Cluster randomized controlled trial
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Masking Description: The single-blind RCT will be applied in the present study, in which the researcher but not the study participants know which intervention has been allocated at the preschool level. In the experimental group, the preschool children will be received the i-MaCHeL program delivers through interactive classroom instruction, and their parents will have access to the i-MaCHeL Web-based program. Whereas in the control group, the preschool children will be received a standard preschool health education curriculum, and their parents will have access to the general Web-based health newsletters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Malaysian Childhood Healthy Lifestyle Program (i-MaCHeL) (Experimental): The preschool children in the experimental group will be exposed to interactive classroom instruction, and their parents will be exposed to the Web-based program. In the experimental group, apart from the standard preschool health education curriculum, the preschool children will also be exposed to the interactive activities and quizzes using Web 2.0 tools, educational videos of a healthy lifestyle, sensory-based food education activities, cooking demonstrations, fun, and active games, and exercises. Whereas the parents will be exposed to Web-based healthy lifestyle educational materials, videos, and pictures sharing, quizzes, and communication through the WhatsApp and closed Facebook groups. Besides, a total of 3 messages per week will be delivered to the parents in the experimental group. The messages will be included announcing the release of a new topic, a reminder to log in to the website and read the health information, and a reminder to participate in the online activities.
  Interventions: Behavioral: Experimental Group: Interactive Malaysian Childhood Healthy Lifestyle Program (i-MaCHeL)
- Standard health education (Active Comparator): The children in the control group do not have exposed to the i-MaCHeL interactive classroom instruction, and their parents do not have access to the i-MaCHeL website materials. Thus, the children will be continued with standard health education only in the preschool setting, and their parents will be received Web-based health newsletters. The Web-based newsletters consist of general health information that are relevant to the preschool life stage. In ensuring that the experimental and control groups appear the same, the topics in the Web-based newsletters will have a look and feel similar nature to the experimental group condition. But still, the topics will not be included the interactive components such as videos and pictures sharing activities, quizzes, individualized feedback, and communication through WhatsApp and closed Facebook groups. Only one message (announcement of the release of a new topic) per week will be delivered to parents of the control group.
  Interventions: Behavioral: Control Group: Standard health education

INTERVENTIONS:
Behavioral: Experimental Group: Interactive Malaysian Childhood Healthy Lifestyle Program (i-MaCHeL) — The preschool children in the experimental group will be received the i-MaCHeL program delivers through interactive classroom instruction, and their parents will have access to the i-MaCHeL Web-based program.
  Arms: Interactive Malaysian Childhood Healthy Lifestyle Program (i-MaCHeL)
Behavioral: Control Group: Standard health education — The children in the control group will be continued with standard health education only in the preschool setting, and their parents will be received general Web-based health newsletters.
  Arms: Standard health education

SUMMARY:
Background: Strategies to treat and prevent obesity are urgently required in Malaysia, and it is now considered a public health priority. Aims: The present study aims to evaluate the effectiveness of the i-MaCHeL intervention for preschool's child-parent dyads. The primary objective of the present study is to compare the changes in the child BMI-for-age z-score at 3- and 9-month after baseline measurement. The secondary objectives of the present study are to compare the changes in child dietary intake, child physical activity, child health-related quality of life, parental self-efficacy, parental role modeling, and parental policies at 3- and 9-month after baseline measurement. Study design: The i-MaCHeL intervention is a single-blind, two-group cluster-randomized controlled trial that evaluates the effectiveness of a 3-month obesity prevention intervention on preschool's child-parent dyads at 3- and 9-month after baseline. The participating preschools (n=12) will be randomized to either the intervention or control group in a 1:1 ratio. The present study will involve 460 child-parent dyads of preschool children aged 5 and 6 years old and their parents in Terengganu, Malaysia. Briefly, the preschool children in the experimental group will be received the i-MaCHeL program delivered through interactive classroom instruction, and their parents will have access to the i-MaCHeL Web-based program. In the control group, the preschool children will be received a standard preschool health education curriculum, and their parents will have access to the general Web-based health newsletters. Instruments: Anthropometric measurements (body weight and height) will be assessed according to the WHO standard procedures. Dietary intake of children will be measured using dietary records for three days. Child physical activity, child health-related quality of life, parental role modeling, parental policies, and parental self-efficacy will be assessed using previously validated parent-proxy questionnaires. Conclusion: The strategies to promote healthy eating in reducing the prevalence of obesity among Malaysian preschool children may have long-term benefits to children's health. The combinations of the two modes of delivery (interactive classroom instruction for preschool children and a Web-based program for parents) will have a strong potential to be effective strategies to sustain child-parent engagement and participation in the health-related behavior change program.

DETAILED DESCRIPTION:
1. Research Hypotheses

   The primary hypothesis of the present study is that the preschool children in the i-MaCHeL intervention group would achieve a significant improvement in BMI z-score compared with those in the comparison group at 3- and 9-month after baseline measurement.

   The secondary hypotheses of the present study, as stated below:
   1. Preschool children in the i-MaCHeL intervention group would achieve significant improvements in dietary intake, physical activity, and health-related quality of life compared with those in the comparison group at 3- and 9-month after baseline measurement.
   2. Parents of preschool children in the i-MaCHeL intervention group would achieve significant improvements in parental self-efficacy, parental role modeling, and parental policies compared with those in the comparison group at 3- and 9-month after baseline measurement.
2. Study Location

   Two districts, which are Kuala Terengganu and Kuala Nerus, will be included in this study. These two districts are chosen based on demographic and logistic factors as it is within 35 miles (56 kilometers) of the study center.
3. Reference Population

   The reference population will be based on a sample population drawn from the MOE public preschools in the Terengganu that are registered at the Ministry of Education Malaysia (MOE). There are 307 MOE public preschools with a total of 11,600 children in Terengganu. All children attending MOE public preschool in the Kuala Terengganu and Kuala Nerus districts will be included as the reference population in the present study.
4. Source Population

   The primary sample consists of 5- and 6-year-olds children (born in the year of 2016 and 2017) that attending MOE public preschools, and their parents, living in the Kuala Terengganu and Kuala Nerus districts. There are 71 MOE public preschools in Kuala Terengganu (n=45 preschools) and Kuala Nerus (n=26 preschools), with a total of 1,850 and 1,175 children, respectively.
5. Study Participants

   The preschool's child-parent dyads that fulfill the selection criteria of the present study will be eligible for inclusion. In total, 12 preschools with 460 child-parent dyads will be recruited.
6. Sample Size Determination

   The present study is a preschool-based cluster-randomized controlled trial that evaluates the effectiveness of a 3-month obesity prevention intervention in preschool's child-parent dyads. Twelve preschools with approximately 38 child-parent dyads per preschool, will be enrolled in the present study at baseline. With at least 90% power to identify a small to medium effect size at the 5% significance level, the present study needs a sample of size 460 child-parent dyads. The intervention and control group will each have 230 child-parent dyads in the sample.
7. Sampling Frame

   All preschools located in the Kuala Terengganu and Kuala Nerus districts (n=71), with a total of 3,025 children, will be assessed for inclusion. The preschools with fewer than 38 children (minimum cluster size) or preschools with "special measures" (unlikely to have the capacity to contribute to the study) will be excluded from the study. After the inclusion and exclusion criteria screening, a list of 37 preschools (n= 1,850 children) will be expected to be eligible and invited to participate in the present study. From the list, only 12 preschools will be recruited in the study. The list of all children attending the included preschools will be obtained from the preschool teachers.
8. Sampling Method

   A cluster random sampling technique (probability sampling) at the preschool level will be conducted in the present study. Thirty-seven preschools (expected to be eligible) will be randomly ordered using a random number generator to generate a list of random numbers, and sequentially will be invited to participate. All the preschools will be contacted, and 12 of them will be recruited in the study.
9. Randomization

   Notably, the randomization into intervention and control groups will only occur at the preschool level. Thus, randomization will be carried out at the preschool level rather than the child participants level to minimize the possibility of the experimental group participants would influence by the participants in the control group. In total, 12 preschools, 6 per arm, will be randomized into either the experimental or control group in a 1:1 ratio. After the baseline measures are completed, the participating preschools will be randomized at the start of the preschool year using a randomization computer program of Research Randomizer (version 4.0). The data analyst who randomized the preschools has no contact with the principal researcher, preschool personnel, or study participants.
10. Overview of the Interactive Malaysian Childhood Healthy Lifestyle Program (i-MaCHeL) intervention

    The i-MaCHeL intervention is designed in an innovative approach to delivering a health-related behavior change program among preschool's child-parent dyads to prevent childhood obesity. The i-MaCHeL intervention encourages children to practice a healthy lifestyle and educate parents to shape home lifestyles for optimal child growth and development. Furthermore, the i-MaCHeL intervention is unique, given its Web-based approach to enhance the tool's adoption with hard-to-reach populations, contributing to the long-term goal for childhood obesity prevention. The combinations of the two modes of delivery (interactive classroom instruction for preschool children and a Web-based program for parents) will have a strong potential to be effective strategies to sustain child-parent engagement and participation in the health-related behavior change program.

    In recognition of the value of multiple theoretical approaches, the strong theoretical basis consists of Social Cognitive Theory (SCT), Health Belief Model (HBM), and Trans-Theoretical Model (TTM) principles will be underpinning the development of the i-MaCHeL intervention. These theories' concepts and principles will be ensured to well suited with the i-MaCHeL in supporting desired healthy lifestyle behaviors and healthier weight outcomes. The main contents of the i-MaCHeL program are healthy eating, active physical activity (moderate-intensity exercise), and sedentary behavior (sleep and screen time), which are based on evidence-based national recommendations for a healthy lifestyle targeting preschool children. Educational and behavior change materials of a healthy lifestyle will be developed by following the guidelines from the Malaysian Dietary Guidelines for Children and Adolescents.
11. Intended Statistical Analysis

Differences in changes over time between the intervention and comparison groups will be assessed for each outcome. General linear model repeated measure analysis will be used to determine differences between groups over time (baseline, 3-month, and 9-month) with adjustment for potential covariates. Intention-to-treat (ITT) principles will be applied for parametric data, with all participants analyzed in both intervention and control groups regardless of whether they attended all data collection time points or completed the intervention. Descriptive statistics will be calculated to describe participants' sociodemographic characteristics and scores for each outcome measure by treatment and control groups at baseline, 3-month, and 9-month. Repeated measures analysis of variance (ANOVA) will be conducted to identify significant differences within-group at 3- and 9-month surveys. Whereas repeated measures Analysis of Covariance (ANCOVA) will be performed to determine significant differences between-group at the 3- and 12-month surveys. The measures analyses will be controlled for covariate variables known to influence the outcome measures (child gender, parent education level, parent aged, and parent income). The significance level will be set at < 0.05. Analyses will be performed using Statistical Package for the Social Science (SPSS; version 25.0).

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, children have to be aged 5- or 6-years Malaysian citizens and attending MOE public preschools in the Kuala Terengganu and Kuala Nerus districts. Besides, the parent/guardian of the preschool children must:

* Could read and understand either English or Malay
* To be aged between 25 to 49 years
* Have regular internet access via a tablet device, mobile phone, or computer/laptop
* Have regular access to a phone with texting capability
* Have WhatsApp and Facebook accounts or agreed to create the accounts
* Comfortable to read/view materials on electronic devices
* Willing to complete all questionnaires with their child throughout the study

Exclusion Criteria:

Child-parent dyads will be excluded if they have the following criteria:

* Children that are taking medications or have a medical condition with the potential to affect the weight or restrict age-appropriate play
* Children that are having conditions that require the restriction of certain foods (e.g., celiac disease or food allergies)
* Parents that are suffering from a severe physical or psychological illness, making the study too demanding for the family

Ages: 5 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 460 (Estimated)
Dates: Start 2022-03-16 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in child BMI-for-age z-score | 3-month and 9-month after baseline
  Anthropometric measurements such as body weight and height will be assessed according to the standard procedures of the World Health Organization (1995). BMI will be calculated using the standard formula (kg/m2). BMI-for-age Z-score curve, according to the WHO references will be used to classify weight status. The child weight status will be categorized into four categories which are overweight (> +1SD of BMI-for-age z-score), obese (> +2SD of BMI-for-age z-score), thinness/wasting (< -2SD of BMI-for-age z score) and normal weight (+1SD to -2SD of BMI-for-age z-score).

SECONDARY OUTCOMES:
Changes in child dietary intake | 3-month and 9-month after baseline
  Dietary intake information of the children will be obtained from a three-day food record (two weekdays and one weekend) and the average measurement will be taken. A dietary analysis software, Nutritionist Pro Inc. will be used for energy and nutrient analysis.
Changes in child physical activity | 3-month and 9-month after baseline
  Child physical activity duration (including light-, moderate-, and vigorous-intensity) and sedentary behavior (screen time spent in front of a television, computer, tablet, or video game) will be assessed using a validated Preschool-age Physical Activity Questionnaire (Pre-PAQ), a parent-proxy questionnaire. The parents will be required to report on the time spent (in minutes) in the activities their child did "yesterday" and "last weekend". A 3-day mean for the activities will be calculated as an average of one weekday, Saturday, and Sunday. The different kinds of physical activity are categorized into 5 levels: 1. Sedentary - no movement; 2. Sedentary play - limb or trunk moving; 3. Moving slowly; 4. Moving at a moderate pace and; 5. Moving at a fast pace.
Changes in child health-related quality of life (HRQOL) | 3-month and 9-month after baseline
  Child Health-Related Quality of Life (HRQOL) will be assessed using a validated Quality of Life Inventory Version 4.0 (PedsQL) Generic Core Scales, a parent-proxy questionnaire. A 5-point response scale is utilized (0 = never a problem; 4 = always a problem). The Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0) so that a higher score indicates better HRQOL functioning.
Changes in parental self-efficacy | 3-month and 9-month after baseline
  Parental self-efficacy will be assessed using a validated Parental Self-Efficacy for Healthy Dietary and Physical Activity Behaviors in Preschoolers Scale (PDAP), a parent-proxy questionnaire. An 11-point Likert scale will be used to record responses, ranging from 0 (not at all confident) to 10 (completely confident). Twelve of the 21 items from the questionnaire will be summed to yield separate scores for parental self-efficacy for promoting child physical activity, and the other 9 items will be summed to yield scores for parental self-efficacy for promoting child's healthy eating.
Changes in parental role modeling | 3-month and 9-month after baseline
  Parental role modeling will be assessed using a validated Home Environment Survey (HES), a parent-proxy questionnaire. A 5-point Likert scale will be utilized for parental role modeling items with responses ranging from "never" (0) to "always" (4).
Changes in parental policies | 3-month and 9-month after baseline
  Parental policies will be assessed using a validated Home Environment Survey (HES), a parent-proxy questionnaire. A 5-point Likert scale will be utilized for parental policy items with responses ranging from "never" (0) to "always" (4).

CONTACTS AND LOCATIONS:
Overall Officials: AHMAD FAEZI AB.RASHID, Principal Investigator — Universiti Sultan Zainal Abidin
Locations (1):
- Universiti Sultan Zainal Abidin, Kampung Gong Badak, Terengganu, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rashid AFA, Syed Saadun Tarek Wafa SWW, Talib RA, Bakar NMA. Interactive Malaysian Childhood Healthy Lifestyle (i-MaCHeL) programme: a single-arm pilot study. Pilot Feasibility Stud. 2024 May 18;10(1):80. doi: 10.1186/s40814-024-01483-7. PMID 38762727
- [Derived] Rashid AF, Wafa SW, Abd Talib R, Abu Bakar NM. An interactive Malaysian Childhood Healthy Lifestyle (i-MaCHeL) intervention programme to change weight-related behaviour in preschool child-parent dyads: Study protocol of a cluster randomised controlled trial. PLoS One. 2022 Oct 31;17(10):e0276843. doi: 10.1371/journal.pone.0276843. eCollection 2022. PMID 36315523